CLINICAL TRIAL: NCT07347457
Title: Effects of Four Weeks of Functional Rehabilitation on Exercise-induced Hypoalgesia in Individuals With Chronic Low Back Pain: An Exploratory Study
Brief Title: Functional Rehabilitation Effects on Exercise-induced Hypoalgesia in Chronic Low Back Pain
Acronym: ALGO_LC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique de la Mitterie (Other)
Collaborators: Clinique les Peupliers (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-A01049-38; MR-P0006 (Other: Clinique la Mitterie)
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain
Keywords: Chronic Low Back Pain; Functional Rehabilitation; Physical Activity; Exercise-Induced Hypoalgesia
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functional Rehabilitation Program (Experimental): Participants in this arm will undergo a four-week functional rehabilitation program centered on physical activity. The program includes supervised exercise sessions as part of routine rehabilitation care. Participants will complete standardized exercise sessions for assessment purposes during scheduled study visits.
  Interventions: Other: Functional Rehabilitation Program

INTERVENTIONS:
Other: Functional Rehabilitation Program — Program with physical activity as the main component. The program is delivered in a rehabilitation clinic and includes supervised exercise sessions integrated into standard care.

SUMMARY:
Chronic low back pain is a prevalent condition characterized by persistent pain and associated physical and psychosocial limitations. Physical exercise is currently considered a primary treatment to promote positive outcomes in individuals with chronic low back pain. However, pain itself represents a major barrier to regular participation in physical activity.

In healthy individuals, exercise induces hypoalgesia, reflected by an increase in pain detection thresholds following physical activity. Enhancing exercise-induced hypoalgesia may promote adherence to regular physical activity in individuals with chronic low back pain. Previous research suggests that regular physical activity may facilitate exercise-induced hypoalgesia through physiological responses associated with exercise that are influenced by physical activity levels.

Therefore, interventions centered on physical activity may enhance exercise-induced hypoalgesia in individuals with chronic low back pain, potentially contributing to pain reduction and increased engagement in physical activity. The primary objective of this exploratory study is to evaluate the effects of a four-week functional rehabilitation program, with physical activity as its main component, on exercise-induced hypoalgesia in individuals with chronic low back pain

DETAILED DESCRIPTION:
Chronic low back pain is a common condition characterized by persistent and disabling pain located in the lower back, leading to physical and psychosocial limitations in daily life activities. Physical exercise is currently considered the primary therapeutic approach to promote positive outcomes in individuals with chronic low back pain. However, pain itself remains a major barrier to regular and sustained engagement in physical activity in this population.

In healthy individuals, physical exercise induces an analgesic effect known as exercise-induced hypoalgesia, which is reflected by increased pain detection thresholds following exercise. Enhancing exercise-induced hypoalgesia may help improve adherence to regular physical activity among individuals with chronic low back pain. Nevertheless, the mechanisms underlying this phenomenon remain insufficiently understood. Previous research suggests that regular physical activity may facilitate exercise-induced hypoalgesia through physiological responses to exercise that can be modulated by physical activity levels.

Therefore, physical activity-centered rehabilitation programs may enhance exercise-induced hypoalgesia in individuals with chronic low back pain, potentially contributing to pain reduction, increased physical activity participation, and decreased healthcare utilization.

This exploratory, prospective, single-center interventional study aims primarily to evaluate the effects of a four-week functional rehabilitation program, with physical activity as its main component, on exercise-induced hypoalgesia in individuals with chronic low back pain. Exercise-induced hypoalgesia will be assessed by measuring pain detection thresholds before and after a standardized exercise bout using pressure algometry.

Secondary objectives are twofold. First, the study will examine the relationships between exercise-induced hypoalgesia and individual characteristics associated with chronic low back pain, including pain intensity, functional disability, kinesiophobia, hemodynamic responses to exercise, and physical activity level. Second, the study will determine whether changes in exercise-induced hypoalgesia at the end of the rehabilitation program predict the subsequent evolution of pain symptoms, healthcare utilization, and the resumption of daily physical and occupational activities at 3 months, 6 months, and 1 year following the intervention.

Participants aged 18 to 60 years with a diagnosis of chronic low back pain lasting at least three months will be recruited during their admission to a four-week functional rehabilitation program at a single rehabilitation clinic in France. Eligible participants must be able to provide informed consent and have no contraindications to physical activity. Individuals with severe cardiovascular, neurological, or psychiatric disorders, pregnant or breastfeeding women, and individuals with a history of substance abuse will be excluded.

Participants will complete four on-site assessment visits conducted before and during the rehabilitation program, during which pain detection thresholds, questionnaires assessing functional disability and kinesiophobia, physiological responses to exercise, and physical activity levels will be evaluated. Physical activity will be objectively assessed using actimetry. Following completion of the rehabilitation program, participants will be followed longitudinally through telephone interviews conducted at 3 months, 6 months, and 1 year to assess pain evolution, healthcare use, and resumption of daily and professional activities.

The planned sample size is 51 participants, based on previously reported effect sizes for exercise-induced hypoalgesia. The total recruitment period is expected to last up to 24 months, and each participant will be involved in the study for approximately 14 months, including on-site assessments and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participant
* Able to provide written informed consent
* Aged between 18 and 60 years
* Diagnosed with chronic low back pain, defined as persistent low back pain for at least three months
* Enrolled in the functional rehabilitation program at Les Peupliers Clinic
* Affiliated with a health insurance system

Exclusion Criteria:

* Presence of a contraindication to physical activity
* Presence of a severe cardiovascular, neurological, or psychiatric condition
* Pregnant or breastfeeding women
* History of alcohol and/or drug addiction
* Individuals under legal guardianship or curatorship
* Individuals in an emergency situation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-01-07 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pressure pain detection thresholds before and after exercise | Baseline and immediately after exercise during each study visit over the 4-week rehabilitation period
  Pressure pain detection thresholds will be assessed using a handheld pressure algometer. Measurements will be performed at predefined anatomical sites before and immediately after a standardized exercise bout to evaluate exercise-induced hypoalgesia.

SECONDARY OUTCOMES:
Kinesiophobia assessed by the Tampa Scale of kinesiophobia | At baseline and at the end of the 4-week functional rehabilitation program
  Kinesiophobia will be assessed using the Tampa Scale of Kinesiophobia (TSK), a self-reported questionnaire measuring fear of movement and fear of injury related to physical activity. Higher scores indicate greater levels of kinesiophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique les Peupliers, Villeneuve-d'Ascq, France

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and data protection considerations, including the sensitive nature of health-related data and compliance with applicable data protection regulations.